CLINICAL TRIAL: NCT03401567
Title: Effects of Exercises Combined With Blood Flow Restriction on Strength, Joint Position Sense and Functional Motor Performance in Healthy Individuals
Brief Title: Effects of Exercises Combined With Blood Flow Restriction in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Deniz Dere Arasan, Postgraduate Student, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3408-GOA
Record Dates: First submitted 2017-12-23; First posted 2018-01-17 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2017-12

CONDITIONS: Healthy Individuals
Keywords: blood flow restriction; proprioception; functional performance; muscle strength

STUDY DESIGN:
Intervention Model Description: There are 2 groups of 30 people each. Elbow bending exercises with blood flow restriction will be performed to the exercise group during 6 weeks for 3 times a week. Control group will continue daily activities and a brochure on strengthening exercises and protection from injuries.
Who Masked: Participant
Masking Description: All of the participants must have no neck and upper extremity pain, any fracture and surgical history for the upper extremity, cervical and thoracic area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Elbow bending exercises with blood flow restriction will be performed to the exercise group.
  Interventions: Other: Exercise group
- Control group (No Intervention): Control group will continue daily activities and a brochure on strengthening exercises and protection from injuries.

INTERVENTIONS:
Other: Exercise group — Elbow bending exercises with blood flow restriction will be performed to the exercise group during 6 weeks for 3 times a week. The first set of exercises will be 30 repetitions then 3 sets of 15 repetitions. Totally 75 repetitions will be performed. 30 seconds rest interval between sets will be given.
  Arms: Exercise group

SUMMARY:
Purpose of the study is; to investigate the effect of exercises combined with blood flow restriction on strength, proprioception and functional motor performance in healthy individuals. There is no randomized controlled study of the effect of upper extremity exercises performed by restricting blood flow on the joint sensation of individuals and functional motor performance in healthy individuals. For this reason, purpose of the study is; to investigate the effect of exercises combined with blood flow restriction on strength, proprioception and functional motor performance in healthy individuals. Pain intensity with the numerical pain rating scale (NRS), muscle strength with digital hand dynamometer, shoulder and elbow proprioception with inclinometer, functional motor performance with Upper Extremity Closed Kinetic Chain Stabilization Test, Functional Throwing Performance Index, Single Arm Shot Put Test, Modified Pull-Up Test evaluation of 60 healthy individuals without neck and upper extremity pain, the fracture and surgical history for the upper extremity, cervical and thoracic area that prevent them to participate in the study will be made. Participants will randomly be separated into 2 groups of 30 people each. Elbow bending exercises with blood flow restriction will be performed to the exercise group during 6 weeks for 3 times a week accompanied by a physiotherapist. Control group will continue daily activities and a brochure on strengthening exercises and protection from injuries. Evaluations will be repeated 2 times and analyzed before the treatment and at the end of the 6th week. With the project, the investigators aim to improve the strength, improve proprioception and functional motor performance in healthy individuals by performing exercises restricting blood flow. With the achievement of the targets, exercises combined with blood flow restriction can be considered among the treatments protective for injuries, healing proprioception. The investigators also believe that the project will blaze the trail for the studies to be performed on athletes.

DETAILED DESCRIPTION:
Purpose of the study is; to investigate the effect of exercises combined with blood flow restriction on strength, proprioception and functional motor performance in healthy individuals. In recent years, the prevalent blood flow restricting exercises seem to favor the development of skeletal muscles in different populations. Studies show that muscular hypertrophy can be achieved also with low-intensity resistance exercises by restricting blood flow. Moreover, exercises combined with blood flow restriction with low mechanical stress and minimal muscle damage do not require a long regeneration process. In this regard, it is stated that the blood flow restricting exercises have lower risk of injuries than the high intensity resistant exercises. It has been shown that similar positive results can be obtained with low-intensity resistance exercises performed by restricting blood flow with classical strengthening exercises performed without limiting in the muscle cross section area. In addition to strength, proprioception and neuromuscular control is important in individuals' therapeutic benefit rates, skills and functionalities, in returning to sports after sports injuries. The investigators believe that classical strengthening exercises may be a contribution to proprioception and consequently to functional motor performance because of the contribution to the proprioception, the low intensity resistant exercise technique performed by restricting blood flow, as well as providing similar muscle growth muscle growth, being painless and harmless to the musculoskeletal system. In this regard, there is no randomized controlled study of the effect of upper extremity exercises performed by restricting blood flow on the joint sensation of individuals and functional motor performance in healthy individuals. For this reason, purpose of the study is; to investigate the effect of exercises combined with blood flow restriction on strength, proprioception and functional motor performance in healthy individuals. Pain intensity with the numerical pain rating scale (NRS), muscle strength with digital hand dynamometer, shoulder and elbow proprioception with inclinometer, functional motor performance with Upper Extremity Closed Kinetic Chain Stabilization Test, Functional Throwing Performance Index, Single Arm Shot Put Test, Modified Pull-Up Test evaluation of 60 healthy individuals without neck and upper extremity pain, the fracture and surgical history for the upper extremity, cervical and thoracic area that prevent them to participate in the study will be made. Participants will randomly be separated into 2 groups of 30 people each. Elbow bending exercises with blood flow restriction will be performed to the exercise group during 6 weeks for 3 times a week accompanied by a physiotherapist. Control group will continue daily activities and a brochure on strengthening exercises and protection from injuries. Evaluations will be repeated 2 times and analyzed before the treatment and at the end of the 6th week. With the project, the investigators aim to improve the strength, proprioception and functional motor performance in healthy individuals by performing exercises restricting blood flow. With the achievement of the targets, exercises combined with blood flow restriction can be considered among the treatments protective for injuries, healing proprioception. The investigators also believe that the project will blaze the trail for the studies to be performed on athletes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Do not smoke
* Having full range of motion in neck, shoulder, and elbow
* Body mass index (BMI)˂30 kg/m2
* Able to complete the entire study procedure

Exclusion Criteria:

* Having fracture and surgical history for the upper extremity, cervical or thoracic area
* Having any systemic musculoskeletal disease
* Having neck and upper extremity pain
* Having a diagnosis of scoliosis and chest deformity
* Regularly playing sports with overhead activities (tennis, volleyball, handball, etc.)
* Have been exercising regularly for the last 6 months
* A history of anemia
* A history of cerebrovascular disease or myocardial infarction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Strength | Baseline and 6 weeks later
  Change of biceps and triceps muscles strength(in kg, with hand held dynamometer)

SECONDARY OUTCOMES:
Shoulder proprioception | Baseline and 6 weeks later
  Change of shoulder proprioception for three direction: 75 external rotation, 45 internal rotation and 100 abduction (with bubble inclinometer)
Elbow proprioception | Baseline and 6 weeks later
  Change of elbow proprioception for three degrees: 45, 60 and 75 (with digital inclinometer)
Functional motor performance | Baseline and 6 weeks later
  Determine the performance with Upper Extremity Closed Kinetic Chain Stabilization Test (number of touch)
Functional motor performance | Baseline and 6 weeks later
  Determine the performance with Functional Throwing Performance Index (number of correct shots)
Functional motor performance | Baseline and 6 weeks later
  Determine the performance with Single Arm Shot Put Test (distance measurement in cm),
Functional motor performance | Baseline and 6 weeks later
  Determine the performance with Modified Pull-Up Test (number of pulls)

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yesilyaprak SS, Dere D. Elbow flexion training with blood flow restriction improves strength, proprioception, and performance in healthy individuals: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Oct 16;26(1):976. doi: 10.1186/s12891-025-08768-9. PMID 41102692